CLINICAL TRIAL: NCT03055377
Title: N-Acetylcysteine for Youth Cannabis Use Disorder
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Kevin Gray, Professor of Psychiatry and Behavioral Sciences, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pro00054499
Record Dates: First submitted 2017-02-14; First posted 2017-02-16 (Actual); Results first posted 2024-12-17 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-11

CONDITIONS: Cannabis Use Disorder
Keywords: cannabis; marijuana; youth; adolescent; pharmacotherapy; medication; n-acetylcysteine; trial
MeSH Terms: conditions — Marijuana Abuse | interventions — Acetylcysteine

STUDY DESIGN:
Intervention Model Description: 1:1 parallel group allocation randomized placebo controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind placebo-controlled pharmacotherapy trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- N-acetylcysteine (Experimental): N-acetylcysteine 1200 mg twice daily for 12 weeks
  Interventions: Drug: N-acetyl cysteine
- Placebo (Placebo Comparator): Placebo (matched in appearance to N-acetylcysteine to preserve double-blind) twice daily for 12 weeks
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: N-acetyl cysteine — N-acetylcysteine 1200 mg twice daily for 12 weeks (administered orally)
  Arms: N-acetylcysteine
Drug: Placebo oral capsule — Placebo (matched in appearance to N-acetylcysteine to preserve double-blind) twice daily for 12 weeks (administered orally)
  Arms: Placebo

SUMMARY:
This is a 12-week randomized, placebo-controlled trial of N-acetylcysteine for cannabis use disorder (CUD) in youth (N=192). Participants will be randomized to double-blind NAC or PBO, yielding two equally-allocated treatment groups. All participants will receive brief weekly cannabis cessation counseling and medication management. The primary efficacy outcome will be the proportion of negative urine cannabinoid tests during the 12-week active treatment, compared between groups.

DETAILED DESCRIPTION:
Cannabis use is particularly prevalent and problematic among youth. Compared with only one in eleven cannabis-exposed adults, one in six cannabis-exposed youth develops cannabis use disorder. Moreover, youth are more prone than adults to potentially lasting adverse effects of cannabis use, including cognitive impairment, altered brain development, poor educational outcome, and diminished life achievement. Despite this, relatively little work has focused on developing optimally efficacious cannabis use disorder treatments, particularly among youth. Current evidence-based treatments convey generally small to modest effect sizes, and novel approaches are critically needed. Among the most promising approaches is the over-the-counter antioxidant medication N-acetylcysteine (NAC). Our team previously demonstrated superior NAC versus placebo (PBO) abstinence outcomes in youth with CUD who concurrently received the behavioral treatment contingency management (CM). Further work is now needed to test whether NAC is efficacious without a platform of CM. The proposed trial is a 12-week randomized, placebo-controlled trial of N-acetylcysteine for cannabis use disorder (CUD) in youth (N=192). Participants will be randomized to double-blind NAC or PBO, yielding two equally-allocated treatment groups. All participants will receive brief weekly cannabis cessation counseling and medication management. The primary efficacy outcome will be the proportion of negative urine cannabinoid tests during the 12-week active treatment, compared between groups. We will also serially assess cognitive task performance, examining changes in performance among participants who achieve abstinence versus those that do not. This proposed trial is the clear "next step" in the assessment of NAC as an extremely promising youth CUD treatment modality, and is positioned to inform researchers, clinicians, and the general public, addressing a critical need for optimization of youth CUD treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age 14 - 21 years
2. Must be able to understand the study and provide written informed consent (for participants under 18 years old, a parent/legal guardian must be able to provide consent and the participant must be able to provide assent)
3. Must meet current (within last 30 days) DSM-5 criteria for cannabis use disorder
4. Must express interest in treatment for cannabis use disorder
5. Must submit a positive urine cannabinoid test during screening
6. Females must agree to use appropriate birth control methods during study participation: oral contraceptives, contraceptive patch, barrier (diaphragm or condom), levonorgestrel implant, medroxyprogesterone acetate, complete abstinence from sexual intercourse, or hormonal contraceptive vaginal ring

Exclusion Criteria:

1. Allergy or intolerance to N-acetylcysteine
2. Females who are pregnant or lactating
3. Current use of N-acetylcysteine or any supplement containing N-acetylcysteine (must agree not to take any such supplement throughout study participation)
4. Use of carbamazepine or nitroglycerin within 14 days of randomization or expectation of future use during protocol participation
5. Current enrollment in treatment for cannabis use disorder or expectation of other treatment during protocol participation
6. Any use of synthetic cannabinoids (such as K2/Spice) in the 30 days prior to screening or expectation of future use during protocol participation
7. Current moderate or severe substance use disorder, other than cannabis, tobacco, or alcohol
8. Medical history of severe asthma (uncontrolled with medications)
9. History of seizure disorder
10. Any other medical or psychiatric condition or other significant concern that in the Investigator's opinion would impact participant safety or compliance with study instructions, or potentially confound the interpretation of findings

Ages: 14 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 192 (Actual)
Dates: Start 2017-08-03 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-02-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin M Gray, MD, Principal Investigator — Professor of Psychiatry and Behavioral Sciences
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gray KM, Tomko RL, Baker NL, McClure EA, McRae-Clark AL, Squeglia LM. N-acetylcysteine for youth cannabis use disorder: randomized controlled trial main findings. Neuropsychopharmacology. 2025 Apr;50(5):731-738. doi: 10.1038/s41386-025-02061-y. Epub 2025 Feb 5. PMID 39910268

RESULTS

PARTICIPANT FLOW:
Period: Treatment Phase
Arm/Group | N-acetylcysteine | Placebo
Started | 98 | 94
Completed | 70 | 70
Not Completed | 28 | 24
Not completed — Lost to Follow-up | 28 | 24
Period: Post-Treatment Follow-Up
Arm/Group | N-acetylcysteine | Placebo
Started | 70 | 70
Completed | 44 | 49
Not Completed | 26 | 21
Not completed — Lost to Follow-up | 26 | 21

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | N-acetylcysteine | Placebo | Total
Number analyzed (Participants) | 98 | 94 | 192
Age, Continuous [Mean (Standard Deviation); unit: years] | 19.1 (1.3) | 19.2 (1.7) | 19.2 (1.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 46 | 101
  Male | 43 | 48 | 91
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16 | 11 | 27
  Not Hispanic or Latino | 82 | 83 | 165
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 11 | 20
  White | 78 | 73 | 151
  More than one race | 7 | 8 | 15
  Unknown or Not Reported | 3 | 1 | 4
Region of Enrollment [Number; unit: participants]
  United States | 98 | 94 | 192

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Urine Tests With Negative Cannabinoid Results During Treatment
Description: Qualitative urine cannabinoid testing, with cutoff of 50 ng/mL
Time Frame: Weekly urine cannabinoid tests during 12-week active treatment
Population: Enrolled and randomized participants
Measure: Number; unit: Percentage
Units Other Than Participants: Urine cannabinoid tests
Arm/Group | N-acetylcysteine | Placebo
Number analyzed (Participants) | 98 | 94
Number analyzed (Urine cannabinoid tests) | 763 | 785
Percentage | 9.4 | 14.0

ADVERSE EVENTS:
Time Frame: Adverse event data were collected throughout the full 6-month participant enrollment period (includes 12 weeks of study treatment and extended post-treatment follow-up thereafter)
Description: Adverse events were assessed by the medical clinician during participant interviews and coded via MedDRA terminology.
Arm/Group | N-acetylcysteine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/98 | 0/94
Serious Adverse Events (participants affected / at risk) | 0/98 | 0/94
Other Adverse Events (participants affected / at risk) | 86/98 | 73/94
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | N-acetylcysteine (N=98) | Placebo (N=94)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Ear Congestion (Ear and labyrinth disorders) | 2 (2) | 1 (1)
Otitis Media (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Conjunctivitis (Eye disorders) | 1 (1) | 0 (0)
Eyebrow Twitching (Eye disorders) | 1 (1) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 3 (3) | 5 (5)
Decreased Appetite (Gastrointestinal disorders) | 1 (1) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 5 (6) | 8 (8)
Dyspepsia (Gastrointestinal disorders) | 10 (14) | 5 (7)
Flatulence (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastroenteritis (Gastrointestinal disorders) | 5 (5) | 2 (2)
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 14 (16) | 3 (4)
Heartburn (Gastrointestinal disorders) | 3 (3) | 1 (1)
Nausea (Gastrointestinal disorders) | 32 (41) | 16 (22)
Stomachache (Gastrointestinal disorders) | 7 (9) | 4 (5)
Vomiting (Gastrointestinal disorders) | 16 (19) | 9 (12)
Chills (General disorders) | 1 (1) | 0 (0)
Drug Withdrawal Syndrome (General disorders) | 1 (2) | 2 (2)
Early Satiety (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 3 (3) | 2 (2)
Hangover (General disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1)
Tired (General disorders) | 2 (3) | 0 (0)
Chest Pain (General disorders) | 1 (1) | 0 (0)
Allergy to Animals (Immune system disorders) | 0 (0) | 1 (1)
Coronavirus Infection (Infections and infestations) | 1 (1) | 3 (4)
Immunization Reaction (Immune system disorders) | 1 (1) | 0 (0)
Rhinitis Seasonal (Worsening) (Immune system disorders) | 2 (2) | 0 (0)
Abscess (Infections and infestations) | 0 (0) | 1 (1)
Acarodermatitis (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1)
Hordeolum (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 1 (1)
Influenza Like Illness (Infections and infestations) | 2 (2) | 3 (3)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Otitis Media (Infections and infestations) | 0 (0) | 2 (2)
Pharyngitis (Infections and infestations) | 4 (4) | 2 (3)
Pharyngitis Streptococcal (Infections and infestations) | 2 (3) | 0 (0)
Pyrexia (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 5 (7) | 4 (4)
Tinea Cruris (Infections and infestations) | 0 (0) | 1 (1)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 1 (2) | 2 (2)
Viral Upper Respiratory Tract Infection (Infections and infestations) | 23 (30) | 27 (36)
Allergy to arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Animal Bite (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Back Pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Head Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post-traumatic pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Road Traffic Accident (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Sprained Ankle (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Sunburn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Sputum Abnormal (Investigations) | 0 (0) | 1 (1)
Weight Decrease (Investigations) | 1 (1) | 0 (0)
Abnormal Weight Loss (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Decreased Appetite (Metabolism and nutrition disorders) | 9 (9) | 7 (7)
Early Satiety (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Food Intolerance (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Glucose Tolerance Impaired (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Increased Appetite (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint Dislocation (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Joint Stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Limb Injury (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle Weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Neck Swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Plantar Fasciitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 4 (4) | 4 (5)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0)
Dyskinesia (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 25 (30) | 16 (18)
Irritability (Nervous system disorders) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 2 (2) | 0 (0)
Paresthesia (Nervous system disorders) | 0 (0) | 1 (1)
Poor Quality Sleep (Nervous system disorders) | 3 (3) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 1 (1)
Taste Disorder (Nervous system disorders) | 0 (0) | 1 (1)
Abnormal Dreams (Psychiatric disorders) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 1 (2) | 0 (0)
Anxiety (Psychiatric disorders) | 5 (6) | 11 (12)
ADHD (Psychiatric disorders) | 1 (1) | 0 (0)
Depressed Mood (Psychiatric disorders) | 2 (2) | 8 (9)
Hypersomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Increased Suicidal Thoughts (Psychiatric disorders) | 1 (1) | 1 (1)
Insomnia (Psychiatric disorders) | 18 (19) | 14 (14)
Irritability (Psychiatric disorders) | 7 (8) | 5 (5)
Mood Swings (Psychiatric disorders) | 1 (1) | 2 (2)
Nightmares (Psychiatric disorders) | 6 (7) | 4 (4)
Panic Episode (Psychiatric disorders) | 1 (1) | 1 (1)
Vivid Dreams (Psychiatric disorders) | 3 (3) | 3 (3)
Nocturia (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary Tract Infection (Renal and urinary disorders) | 0 (0) | 2 (2)
Dysmenorrhea (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Heavy Menstrual Bleeding (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Polycystic Ovaries (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vulva Cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (9) | 2 (3)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2)
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3)
Throat Irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Viral Upper Respiratory Tract Infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Night Sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (3)
Road Traffic Accident (Social circumstances) | 1 (1) | 0 (0)
Dental Operation (Surgical and medical procedures) | 1 (1) | 1 (1)
Intrauterine Contraception (Surgical and medical procedures) | 1 (1) | 0 (0)
Skin Lesion Removal (Surgical and medical procedures) | 0 (0) | 1 (1)
Hot Flashes (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-14): https://cdn.clinicaltrials.gov/large-docs/77/NCT03055377/Prot_SAP_000.pdf